CLINICAL TRIAL: NCT01822132
Title: Risky Decision Making in Methamphetamine Users: The Role of Opioid Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, P. Todd Korthuis, MD, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ALKIIT-KOR-034; 1R21DA033182-01A1 (NIH)
Record Dates: First submitted 2013-03-21; First posted 2013-04-02 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Methamphetamine Abuse; HIV
MeSH Terms: interventions — vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended release naltrexone (Experimental): One dose of intramuscular injection of 380mg extended-release naltrexone.
  Interventions: Drug: Extended release naltrexone
- Placebo (Placebo Comparator): One dose of intramuscular injection of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extended release naltrexone
  Other Names: Vivitrol
  Arms: Extended release naltrexone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this protocol is to learn more about impulsive decision making in people who use methamphetamines. The investigators would like to know if a medication called naltrexone changes how people make decisions. The investigators would also like to know whether changes in decision making can be observed by MRI (magnetic resonance imaging).

The research is conducted in Portland, OR.

ELIGIBILITY:
Summary Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM)-IV Methamphetamine Dependence
* Deemed healthy enough to participate by study physician
* Age 18-55
* Right handed
* English-speaking

Summary Exclusion Criteria:

* Current opioid use in the last 30 days; opioid abuse or dependence within past 5 years
* Pregnancy
* MRI contraindications (e.g. metal in head).

The research is conducted in Portland, OR.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Korthuis, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon

REFERENCES:
- [Derived] Kohno M, Morales AM, Dennis LE, McCready H, Hoffman WF, Korthuis PT. Effects of Naltrexone on Large-Scale Network Interactions in Methamphetamine Use Disorder. Front Psychiatry. 2019 Sep 3;10:603. doi: 10.3389/fpsyt.2019.00603. eCollection 2019. PMID 31551824
- [Derived] Kohno M, Dennis LE, McCready H, Schwartz DL, Hoffman WF, Korthuis PT. A preliminary randomized clinical trial of naltrexone reduces striatal resting state functional connectivity in people with methamphetamine use disorder. Drug Alcohol Depend. 2018 Nov 1;192:186-192. doi: 10.1016/j.drugalcdep.2018.07.045. Epub 2018 Sep 21. PMID 30266003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After consenting, 13 participants did not meet screening inclusion criteria and were removed from the study and 11 participants withdrew, leaving 52 eligible participants for randomization into a treatment group (Naltrexone or Placebo)
Groups:
- Naltrexone: One dose of intramuscular injection of 380mg extended-release naltrexone.
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 25 | 27
Completed | 21 | 25
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Extended Release Naltrexone: One dose of intramuscular injection of 380mg extended-release naltrexone.
  Extended release naltrexone
- Placebo: One dose of intramuscular injection of placebo.
  Placebo
- Total: Total of all reporting groups
Arm/Group | Extended Release Naltrexone | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 23 | 25 | 48
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Discounting Tasks: Sexual Probability Discounting (SexPD)
Description: In the SexPD task, subjects are asked to choose between having sex with a more appealing partner with a varying chance of having a sexually transmitted infection (STI) or a less appealing partner with no STI.
  A hyperbolic decay model was used to calculate h, a free parameter that indexes the rate of probabilistic discounting. Smaller h values indicate a preference for probabilistic (i.e., riskier) outcomes. To normalize the data, the natural log of h values were calculated and reported here.
Time Frame: 28 days post drug intervention
Population: Subjects with methamphetamine dependence and either HIV positive or not, all abstaining from opioids for at least 30 days.
Measure: Mean (Standard Deviation); unit: natural log
Groups:
- Naltrexone: Participants who were randomized to naltrexone.
- Placebo: Participants who were randomized to receive placebo.
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 21 | 25
natural log
  Baseline_All | 2.97 (11.07) | 6.52 (8.52)
  Post_All | 4.68 (12.07) | 7.67 (11.74)
  Post_HIV-positive: number analyzed (Participants) | 6 | 6
  Post_HIV-positive | -0.54 (5.16) | 1.08 (2.84)
  Post_HIV-negative: number analyzed (Participants) | 15 | 19
  Post_HIV-negative | 6.55 (13.39) | 9.79 (13.38)

2. Primary Outcome: Discounting Tasks: Standard Delay Discounting (DD)
Description: Monetary delay discounting task consisted of choosing between a larger, delayed and a smaller, immediate reward. A hyperbolic decay model was used to calculate k, a free parameter that indexes the rate of delay discounting. As k values are typically skewed across subjects, the distribution of k was normalized by using a natural log transformation. The normalized values are reported here. If k typically ranges between 0.5 and 10^-5, then the natural log of k will range between -0.69 and -11.5. Larger normalized k values indicate a preference for smaller sooner outcomes (i.e., more impulsive decision-making).
Time Frame: 28 days post drug intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: natural log
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 21 | 25
natural log
  Baseline_All | -2.92 (6.06) | -3.90 (2.04)
  Post_All | -2.73 (7.76) | -4.25 (1.65)
  Post_HIV-positive | -5.44 (1.48) | -5.56 (1.61)
  Post_HIV-negative | -1.57 (9.08) | -3.88 (1.50)

3. Primary Outcome: Barrat Impulsiveness Scale (BIS)
Description: The Barrat Impulsiveness Scale (BIS) is a 30 item questionnaire to measure a persons impulsiveness. Items are answered on a 4-point scale and scored 1-4 then summed across responses. Total scores range from 30-120 with a higher summed score indicating higher impulsivity.
Time Frame: 28 days post drug intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Naltrexone: Participants randomized to naltrexone.
- Placebo: Participants randomized to placebo.
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 21 | 25
score on a scale
  Baseline_All | 77.5 (14.24) | 73.52 (13.16)
  Post_All | 71.79 (10.07) | 63.30 (11.53)
  Post_HIV-positive: number analyzed (Participants) | 6 | 6
  Post_HIV-positive | 70.83 (7.49) | 61 (13.15)
  Post_HIV-negative: number analyzed (Participants) | 15 | 19
  Post_HIV-negative | 72.23 (11.31) | 64.47 (11.70)

4. Primary Outcome: Risk Assessment Battery (RAB)
Description: The Risk Assessment Battery (RAB) is a 26 question self-administered assessment focusing on drug use, injection and sexual risk during the past 30 days.
  Three composite HIV risk scores (drug, sex, and total score) are calculated. The questions have different numbers of items, and scores for a single question can range from 0 to 7, with higher values reflecting more instances of risk behavior. The drug risk score has a range of 0 to 22 and is calculated from 8 questions that address recent substance use, including frequency, needle sharing, and cleaning of the "works." 9 questions are used to calculate a sex risk score that has a range of 0 to 18, and these questions address the frequency and types of sexual behavior, HIV status of sexual partners, and type of protection that was used (if any). Total score is calculated by adding drug and sex scores and dividing by 40, the maximum score possible, and ranges from 0 to 40 where higher scores indicate greater risk behavior.
Time Frame: 28 days post drug intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 21 | 25
score on a scale
  DrugRisk_Baseline_All | 1.33 (2.92) | 0.6 (1.87)
  DrugRisk_Post_All | 0.24 (0.54) | 0.08 (0.40)
  SexRisk_Baseline_All | 5.48 (3.23) | 4.44 (3.16)
  SexRisk_Post_All | 4.81 (2.75) | 4.72 (2.89)
  TotalRisk_Baseline_All | 0.17 (0.12) | 0.13 (0.09)
  TotalRisk_Post_All | 0.13 (0.07) | 0.12 (0.07)
  DrugRisk_Baseline_HIV-positive: number analyzed (Participants) | 6 | 6
  DrugRisk_Baseline_HIV-positive | 1 (1.67) | 0.17 (0.41)
  DrugRisk_Post_HIV-positive: number analyzed (Participants) | 6 | 6
  DrugRisk_Post_HIV-positive | 0 (0) | 0 (0)
  SexRisk_Baseline_HIV-positive: number analyzed (Participants) | 6 | 6
  SexRisk_Baseline_HIV-positive | 6.5 (4.04) | 5.17 (2.64)
  SexRisk_Post_HIV-positive: number analyzed (Participants) | 6 | 6
  SexRisk_Post_HIV-positive | 5.83 (3.76) | 4.17 (1.83)
  TotalRisk_Baseline_HIV-positive: number analyzed (Participants) | 6 | 6
  TotalRisk_Baseline_HIV-positive | 0.19 (0.08) | 0.13 (0.06)
  TotalRisk_Post_HIV-positive: number analyzed (Participants) | 6 | 6
  TotalRisk_Post_HIV-positive | 0.15 (0.094) | 0.10 (0.05)
  DrugRisk_Baseline_HIV-negative: number analyzed (Participants) | 15 | 19
  DrugRisk_Baseline_HIV-negative | 1.47 (3.34) | 0.74 (2.13)
  DrugRisk_Post_HIV-negative: number analyzed (Participants) | 15 | 19
  DrugRisk_Post_HIV-negative | 0.33 (0.62) | 0.11 (0.46)
  SexRisk_Baseline_HIV-negative: number analyzed (Participants) | 15 | 19
  SexRisk_Baseline_HIV-negative | 5.07 (2.91) | 4.21 (3.34)
  SexRisk_Post_HIV-negative: number analyzed (Participants) | 15 | 19
  SexRisk_Post_HIV-negative | 4.4 (2.26) | 4.89 (3.18)
  TotalRisk_Baseline_HIV-negative: number analyzed (Participants) | 15 | 19
  TotalRisk_Baseline_HIV-negative | 0.16 (0.13) | 0.12 (0.095)
  TotalRisk_Post_HIV-negative: number analyzed (Participants) | 15 | 19
  TotalRisk_Post_HIV-negative | 0.12 (0.055) | 0.13 (0.081)

5. Secondary Outcome: Methamphetamine Use
Description: Participants were asked "How many days in the past 30 days did you use methamphetamine?". This is a self-report measure.
Time Frame: 28 days post drug intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Extended Release Naltrexone | Placebo
Number analyzed (Participants) | 21 | 25
days
  Post_All | 1.33 (3.23) | 2.17 (5.52)
  Post_HIV-positive | 1.17 (1.83) | 1.6 (3.58)
  Post_HIV-negative | 1.4 (3.70) | 0.13 (0.52)

ADVERSE EVENTS:
Arm/Group | Extended Release Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No